CLINICAL TRIAL: NCT03225651
Title: Autologous Bone Marrow Stem Cell Therapy Combined With Psychological Therapy and Rehabilitation for Autism: An Open Label Controlled Clinical Trial
Brief Title: Autologous Bone Marrow Stem Cell Therapy Combined With Psychological Therapy and Rehabilitation for Autism
Acronym: ASPRA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vinmec Research Institute of Stem Cell and Gene Technology (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VinmecRISCGT69
Record Dates: First submitted 2017-07-05; First posted 2017-07-21 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2018-11

CONDITIONS: Stem Cell Transplantation
Keywords: Stem cell; Autism; Psychological; Rehabilitation
MeSH Terms: conditions — Autistic Disorder | interventions — Stem Cell Transplantation; Rehabilitation

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stem cell transplantation (Experimental): Stem cell transplantation 2 intrathecal administrations of autologous bone marrow mononuclear cells at baseline and 6 months afterward
  Interventions: Biological: Stem cell transplantation; Behavioral: Psychological therapy and Rehabilitation
- Psychological therapy and rehabilitation (Experimental): Psychological therapy Rehabilitation in 3 months
  Interventions: Biological: Stem cell transplantation; Behavioral: Psychological therapy and Rehabilitation

INTERVENTIONS:
Biological: Stem cell transplantation — Transplantation of Autologous Bone Marrow Mononuclear cells
Behavioral: Psychological therapy and Rehabilitation — Psychological Therapy and Rehabilitation for autism children around 3 months

SUMMARY:
The aim of this study was to evaluate the safety and effectiveness of autologous bone marrow mononuclear stem cells combined with Psychological Therapy and Rehabilitation for Autism children

DETAILED DESCRIPTION:
The aim of this study was to evaluate the safety and effectiveness of autologous bone marrow mononuclear stem cells combined with Psychological Therapy and Rehabilitation in the management of autism of 60 patients at Vinmec Research Institute of Stem Cell and Gene Technology Hanoi, Vietnam from January 2017 to December 2018

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of autism according to the Diagnostic and Statistical Manual-V diagnostic criteria for autistic disorder

Exclusion Criteria:

* Epilepsy
* Hydrocephalus with ventricular drain
* Coagulation disorders
* Allergy to anesthetic agents
* Severe health conditions such as cancer, failure of heart, lung, liver or kidney
* Active infections
* Severe psychiatric disorders
* Rett syndrome
* Fragile X syndrome

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2017-07-18 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Assess the change in autism level by using tools | 6 months and 12 months after transplantation
  using total score of childhood autism rating scale, autism diagnostic observation schedule second edition, DENVER II, Indian Scale for assessment of Autism
Evaluate the safety of therapy by record number of adverse events | Through study completion, an average of 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Vinmec Research Institute of Stem Cell and Gene Technology, Hanoi, Vietnam

REFERENCES:
- [Derived] Than UTT, Nguyen LT, Nguyen PH, Nguyen XH, Trinh DP, Hoang DH, Nguyen PAT, Dang VD. Inflammatory mediators drive neuroinflammation in autism spectrum disorder and cerebral palsy. Sci Rep. 2023 Dec 18;13(1):22587. doi: 10.1038/s41598-023-49902-8. PMID 38114596
- [Derived] Nguyen Thanh L, Nguyen HP, Ngo MD, Bui VA, Dam PTM, Bui HTP, Ngo DV, Tran KT, Dang TTT, Duong BD, Nguyen PAT, Forsyth N, Heke M. Outcomes of bone marrow mononuclear cell transplantation combined with interventional education for autism spectrum disorder. Stem Cells Transl Med. 2021 Jan;10(1):14-26. doi: 10.1002/sctm.20-0102. Epub 2020 Sep 9. PMID 32902182